CLINICAL TRIAL: NCT00665600
Title: A Double-Blind, Randomized, Multicenter, Parallel-Group Study of Levalbuterol in the Treatment of Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Safety of Levalbuterol in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 051-914
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Chronic Bronchitis; Chronic Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Levalbuterol 0.63 mg TID
  Interventions: Drug: Levalbuterol HCl
- 2 (Experimental): Levalbuterol 1.25 mg TID
  Interventions: Drug: Levalbuterol HCl
- 3 (Active Comparator): Racemic Albuterol 2.5 mg TID
  Interventions: Drug: Albuterol Sulfate
- 4 (Placebo Comparator): Placebo TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levalbuterol HCl — Levalbuterol 0.63 TID
  Other Names: Xopenex HCl Inhalation Solution
  Arms: 1
Drug: Levalbuterol HCl — Levabuterol 1.25 mg TID
  Other Names: Xopenex HCl Inhalation Solution
  Arms: 2
Drug: Albuterol Sulfate — Racemic albuterol 2.5 mg TID
  Other Names: Ventolin Inhalation Solution
  Arms: 3
Drug: Placebo — Placebo TID
  Arms: 4

SUMMARY:
To investigate the efficacy and safety of repeated dosing of Levalbuterol over 6 weeks of treatment in COPD.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, double-blind, placebo and active controlled, parallel-group study of adult subjects with COPD. Approximately 250 subjects will be enrolled to randomize at least 200 subjects. Study participation will consist of a total of six study visits over nine weeks for each subject. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must be at least greater than or equal to 35 years of age at the time of consent.
* Subjects must have a pre-established primary clinical diagnosis of COPD.
* Subjects must have a baseline FEV1 less than or equal to 65%
* Subjects must have a predicted and >0.70 Liter
* subject was taking steroids (inhaled, oral, or nasal), short-acting xanthines, or leukotrienes, the dose must have been stable for 30 days
* Subjects must have a FEV1/forced vital capacity (FVC) less than or equal to 70%
* Subjects must have a greater than or equal to 15 pack-year smoking history
* Subjects must have a baseline medical research council (MRC) dyspnea scale score greater than or equal to 2
* Regular use of a prescribed therapy for control of COPD symptoms for 3 months prior to study entry.
* No COPD exacerbations that have required an emergency room visit, hospital admission or intensive out-patient therapy within 1 month prior to study entry

Exclusion Criteria:

* Females who are pregnant or lactating.
* Concurrent requirement of oxygen therapy
* Known history of asthma, or any chronic respiratory disease other than COPD (not including chronic bronchitis or emphysema).
* Diagnosis of cancer within 5 years prior to study entry with the exception of non-melanoma skin cancer.
* Lung resection of more than one full lobe.
* Use of intravenous, intra-articular or intramuscular corticosteroids within 30 days of study entry
* History of upper or lower respiratory infection within 14 days of study entry.
* Participation in an investigational drug study within 30 days of study entry.

Ages: 35 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2002-02; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the time-normalized area under the percent change from visit predose in FEV1 curve (nAUC0-8 hours) averaged over the six week double-blind period. | Days -21, -14, 0, 14, 28, and 42

SECONDARY OUTCOMES:
Spirometry parameters | Days -21, -14, 0, 14, 28, and 42
Exacerbations of COPD | Days -14, 0, 14, 28, 42
COPD symptom ratings | Days 0, 14, 28, 42
Baseline dyspnea and transitional dyspnea indices | Days 0, 14, 28, 42
Ipatropium Bromide MDI use | Day 0, 14, 28, 42
Short acting Beta-agonist MDI use | Days 0, 14, 28, 42
Subject and physician global evaluations | Days 14, 28, 42
St. George's Hospital Respiratory Questionnaire (SGRQ). | Days 0, 42

CONTACTS AND LOCATIONS:
Locations (24):
- United States (20):
  - Carmichael, California
  - Spring Valley, California
  - Wheat Ridge, Colorado
  - Largo, Florida
  - Miami, Florida
  - Panama City, Florida
  - Atlanta, Georgia
  - Elk Grove Village, Illinois
  - Hines, Illinois
  - Wheaton, Maryland
  - Springfield, Massachusetts
  - Cadillac, Michigan
  - Columbia, Missouri
  - Missoula, Montana
  - Springfield, New Jersey
  - Chapel Hill, North Carolina
  - Mogadore, Ohio
  - Providence, Rhode Island
  - Austin, Texas
  - San Antonio, Texas
- Canada (4):
  - Calgary, Alberta
  - Winnepeg, Manitoba
  - Mississauga, Ontario
  - Toronto, Ontario